CLINICAL TRIAL: NCT01345422
Title: A Pilot Study to Assess the Usefulness of the Wii Balance Board for Dizziness
Brief Title: Wii Balance Board in Dizziness
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study never started since it did not receive IRB approval
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HNS1
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Dizziness
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Wii Balance Board (Experimental): Wii Balance Board Training
  Interventions: Other: Wii Balance Board

INTERVENTIONS:
Other: Wii Balance Board — Participant will undergo Nintendo Wii Balance Board training for two months , five days a week for 30 minutes

SUMMARY:
Patients with dizziness presently undergo physical therapy rehabilitation. Our study will study whether Wii Balance Board made by Nintendo Inc. will be helpful in patients with dizziness. They will undergo dizziness evaluation to quantify their dizziness.

ELIGIBILITY:
Inclusion Criteria:

* Abnormal posturography exam

Exclusion Criteria:

* Pregnant Women and children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Cheng, MD, Principal Investigator — Southern California Permanente Medical Group

IPD SHARING:
Plan to Share IPD: No
this study did not receive IRB approval